CLINICAL TRIAL: NCT00213304
Title: Safety and Immunogenicity of Live Attenuated Oka/Merck Varicella Vaccine in Children Listed to Undergo Solid Organ Transplantation
Brief Title: The Safety of Oka Varicella in Children Prior to Solid Organ Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Upton Allen, Chief, Division of Infectious Diseases, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0019990029
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Organ Transplantation; Immunosuppression
Keywords: organ transplantation; immunosuppression; vaccine; varicella; pediatrics
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

ARMS (1):
- varicella vaccine (VARIVAX) (Experimental): varicella vaccine (VARIVAX)
  Interventions: Biological: varicella vaccine (VARIVAX)

INTERVENTIONS:
Biological: varicella vaccine (VARIVAX)

SUMMARY:
This study sought to determine the safety of the varicella vaccine pre- and post-transplantation when given to pediatric patients listed for solid organ transplantation. The study assessed the antibody response to a two-dose vaccine regimen and determined the durability of that antibody response at several intervals in the post-transplant period. As a secondary objective, the relationship between antibody titers and different variables were explored

ELIGIBILITY:
Inclusion Criteria:

* Children > 9 months of age and adolescents < 18 years of age.
* Pediatric transplant candidates who are in any of the following categories:

  1. listed to receive kidney, liver, heart, lung or other or solid organ transplantation in a Canadian transplant centre
  2. not yet officially listed, but are regarded by their physicians as transplant candidates by virtue of their underlying diseases
* No clinical history for varicella.
* Seronegative for antibodies to VZV except infants 9 - 12 months of age who may be seropositive due to maternal antibodies.
* Informed consent obtained

Exclusion Criteria:

* Previous immunization with varicella vaccine.
* Any established immune deficiency (underlying disease or drug induced) or any neoplastic disease
* Children on any oral and / or intravenous steroids within 3 months prior to immunization. Children on inhaled corticosteroids in excess of 800 mcg of beclomethasone dipropionate ( or equivalent ) per day.
* Any exposure to varicella or herpes zoster in the previous 4 weeks involving household, playmate or hospital contacts.
* Inability to delay the transplantation for up to 6 weeks following the last varicella immunization.
* Presence of a person at increased risk for varicella infection in direct and unavoidable proximity with the vaccinees ( e.g. an immunocompromised sibling)
* Past history of varicella or known positive antibody titer for varicella except infants 9 - 12 months of ages who may be seropositive due to maternal antibodies
* Known hypersensitivity to any of the components of the vaccine, including neomycin and gelatin
* Patients whose mothers are known to be seronegative and plan to become pregnant in the subsequent three months
* Administration of VZIG or any other blood products in the previous six weeks (packed red blood cells excepted).
* Any significant infection and/or fever at the time of vaccination
* Any patient receiving or planning to receive salicylates in the six weeks after immunization
* Any patient who has received any live vaccine for 6 weeks or killed vaccine for 2 weeks prior to or after the scheduled VARIVAX™ vaccination.

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 1999-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Determination of the safety of VARIVAX™ | Up to 6 months
  Eligible subjects given a two-dose OMVV pre transplantation were monitored for Adverse Events. AE were monitored for up to six wk after each dose with the assistance of parent diaries.
Determination of the safety of VARIVAX™ | up to 6 months
  All transplant recipients were monitored over the follow-up period for microbiological and clinical evidence of reactivation of other herpes group viruses.
Determination of the proportion immunized who demonstrate seroconversion and maintain humoral immunity seroconversion at 6, 12 and 24 months post-transplantation | up to 12 months
  Control antigen was prepared in parallel from uninfected cells. A gpELISA antibody level of >0.6 gpEU/mL defined seroconversion, and a gpELISA antibody level exceeding 5 gpEU/mL defined seroprotection.
Determination of the proportion immunized who demonstrate seroconversion and maintain humoral immunity seroconversion at 6, and 12 months post-transplantation | Up to 12 months
  VZV-specific antibodies were measured at Merck Research Laboratories using a previously validated ELISA method that detected antibodies to VZV glycoproteins purified from VZV-infected human fibroblasts.

CONTACTS AND LOCATIONS:
Overall Officials: Upton Allen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada; Upton Allen, Study Chair — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada